CLINICAL TRIAL: NCT00974779
Title: Application of the "High-cutoff (HCO1100)" Hemodialyzer to Reduce Chronic Inflammation in Hemodialysis Patients With Elevated CRP Levels
Brief Title: High-cutoff Hemodialyzer to Reduce Chronic Inflammation in Hemodialysis Patients
Acronym: HCO1100
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Gambro Dialysatoren GmbH (Industry); KfH Kuratorium für Dialyse und Nierentransplantation e.V., Neu Isenburg, Germany (Unknown)
Responsible Party: Principal Investigator, Matthias Girndt, Professor of Internal Medicine, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KIM2H-2009-02
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: End Stage Renal Disease
Keywords: kidney failure chronic; renal dialysis; inflammation; monocytes; end stage renal disease on regular thrice weekly hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HCO dialyzer (Experimental): Hemodialysis with the HCO1100 hemodialyzer membrane with high molecular weight cut off.
  Interventions: Device: HCO1100 dialyzer
- Placebo (Active Comparator): Regular dialysis using a polyamide high-flux hemodialyzer
  Interventions: Device: regular dialysis polyamide

INTERVENTIONS:
Device: HCO1100 dialyzer — Thrice weekly dialysis using the HCO1100 dialyzer for 4.5h, 2 weeks
  Other Names: Gambro HCO1100
  Arms: HCO dialyzer
Device: regular dialysis polyamide — Continuation of the regular hemodialysis using polyamide high-flux hemodialysers
  Other Names: Gambro Polyflux 11
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether a dialyzer with a higher than usual permeability for proteins can eliminate proinflammatory proteins from the blood of patients on regular maintenance hemodialysis who have chronically elevated levels of inflammation markers such as C-reactive protein (CRP) in their blood.

DETAILED DESCRIPTION:
Patients with ESRD on chronic hemodialysis patients frequently have elevated markers of inflammation (e.g. serum CRP values). Hemodialysis may clear the blood from low molecular weight toxins and retention products such as creatinine, potassium, or urea. The dialyzer clearance of middle to high molecular weight substances such as cytokines and cytokine receptors is low. Nearly 50% of chronic dialysis patients have persistent subclinical inflammation which is strongly associated with cardiovascular disease and mortality. The study tests the hypothesis that removal of proteins in the weight range of 10.000-30.000 D via a more permeable dialyzer membrane reduces chronic inflammation in these patients.

ELIGIBILITY:
Inclusion Criteria:

* regular hemodialysis for at least 3 months
* treatment thrice weekly
* high-flux hemodialyzer for at least 4 weeks
* age > 18 years and < 80 years
* at least one CRP value > 5mg/L within 8 weeks before inclusion
* able to understand and consent the study
* written informed consent

Exclusion Criteria:

* no consent
* clinically apparent acute infection
* CRP > 50 mg/L
* serum albumin < 3,5 mg/L
* central venous line as dialysis access
* immunosuppressive medication
* pregnancy or lactation
* inclusion into any other interventional trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Inflammation: CRP plasma level and quantity of circulating CD14/16 positive monocytes | 2 weeks

SECONDARY OUTCOMES:
Serum albumin losses | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine II, Martin-Luther-University Medical School, Halle, Saxony-Anhalt, Germany

REFERENCES:
- [Derived] Fiedler R, Neugebauer F, Ulrich C, Wienke A, Gromann C, Storr M, Bohler T, Seibert E, Girndt M. Randomized controlled pilot study of 2 weeks' treatment with high cutoff membrane for hemodialysis patients with elevated C-reactive protein. Artif Organs. 2012 Oct;36(10):886-93. doi: 10.1111/j.1525-1594.2012.01479.x. Epub 2012 Jul 30. PMID 22845695